CLINICAL TRIAL: NCT02498847
Title: Occupational Therapy-Delivered Cognitive Behavioral Therapy for Symptomatic Knee Osteoarthritis: A Pilot Study
Brief Title: Occupational Therapy-Delivered Cognitive Behavioral Therapy for Symptomatic Knee Osteoarthritis
Acronym: ENGAGE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00067979
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — engage 8200

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ENGAGE intervention (Experimental): 8 in-person weekly treatment sessions with an occupational therapist of 30 minutes - 1 hour duration intervention content provided on website, homework assigned each week after intervention period, monthly calls conducted to check on health status
  Interventions: Behavioral: ENGAGE
- Usual Care (No Intervention): participated in usual care and received monthly calls to check on health status

INTERVENTIONS:
Behavioral: ENGAGE — Participants are introduced to ENGAGE program by the study OT. The ENGAGE program is located on a website and has several modules. The modules include a video in which a health provider is featured. This health provider gives a short presentation on a topic related to OA, symptom management or lifestyle change. Within each module, there is downloadable homework and additional information which can be printed. The modules are:
  * What is Osteoarthritis?
  * Information about treatments
  * Exercise
  * Sleep hygiene
  * Relaxation
  * Pleasant Activity Scheduling
  * Goal setting
  * Problem Solving
  * Pacing
  * Communication
  Arms: ENGAGE intervention

SUMMARY:
Knee osteoarthritis (OA) affects 27 million US adults and is a leading cause of pain and disability. Non-pharmacological interventions are recommended but are underutilized. Exercise reduces pain and improves physical function, but benefits tend to wane without a component to facilitate behavior change. Cognitive behavioral therapy (CBT) has long term benefits on pain and physical function in individuals with OA, but is not typically offered in clinical care. CBT could be taught in the context of clinical care by occupational therapists (OT). OTs help people manage chronic conditions by teaching behavioral strategies that promote health and function. The purpose of this study is to test the feasibility and efficacy of an OT-delivered cognitive behavioral therapy program to help people manage their knee OA.

DETAILED DESCRIPTION:
Knee OA, in particular, is a major driver of health care costs and is also a leading cause of arthritis-related activity limitations. A common assumption in knee OA treatment is that relief of joint pain will lead to improvements in physical function. However, many factors can influence disability in OA, not only the biomechanical factors which have been the focus of traditional rehabilitation. Although research supports a broader biopsychosocial approach to knee OA treatment, it has not been broadly adopted into clinical treatments. The biopsychosocial model posits that pain and disability are not only affected by pathophysical (e.g., biological) factors, but also psychological (e.g., depression, coping, self-efficacy) and social factors (e.g., social support, response of significant other).

One approach to offering psychosocial aspects in the context of pain treatment has been via CBT, a common psychosocial intervention, with evidence supporting its efficacy in OA. Despite the evidence, CBT is rarely integrated into actual clinical practice for people with knee OA. Barriers to integration have included limited access to psychologists (particularly in rural settings), difficulties coordinating primary care physicians with psychological practices, inconsistent reimbursement of psychological services for OA pain, and inconsistent standardization of treatments across settings. The current study aims to overcome barriers that have previously limited access to a biopsychosocial approach to knee OA treatments by integrating cognitive and behaviorally-based self-management training into a new rehabilitation intervention offered through occupational therapy, an allied medical field which commonly teaches behavioral strategies to improve physical function in many clinical populations. Because this approach will be manualized, it will provide the opportunity for easy adoption into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* community-living
* report of at least mild to moderate pain in knee with osteoarthritis
* clinical determination of knee osteoarthritis
* report of knee pain for > 3 months duration
* ambulatory with or without cane or walker
* has internet access and can use computer

Exclusion Criteria:

* severe physical impairment
* current cancer treatment
* knee injections or surgery in previous 3 months
* using long-acting narcotics
* shift workers
* participation in rehabilitation or behavioral therapy for OA in the previous year

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Self-Reported Physical Function-WOMAC | 5 minutes
  Western Ontario and McMaster University Arthritis Index (WOMAC) 17 items, participants rate difficulty in performing different activities on a 0 - 4 scale

SECONDARY OUTCOMES:
Objective Physical Function- 6 minute walk test | 6 minutes
  The 6 minute walk test involves walking at usual pace for 6 minutes over a flat surface. Overall distance is recorded (in feet).
Pain - Brief Pain Inventory | 5 minutes
  10 item scale in which participants report their pain severity and interference on a 0 - 10 scale
Patient Global Impression of Change | <5 minutes
  Participant answers one question. Overall how do you feel since you started participating in this study? on a scale of very much improved (1) - very much worse (7)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Murphy, ScD OTR, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - University of Michigan Institute of Gerontology, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan